CLINICAL TRIAL: NCT04305509
Title: Outcomes After Chiropractic Spinal Manipulative Therapy for Patients With Lumbar Disc Herniation and Radiculopathy
Brief Title: Outcomes After Chiropractic Spinal Manipulative Therapy With Lumbar Disc Herniation and Radiculopathy
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Brigitte Wirth, Senior scientist Chiropractic Medicine, Balgrist University Hospital
Other Study IDs: PB_2019_00151
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Lumbar Disc Herniation
Keywords: long-term outcome
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LDH patients: Patients with lumbar disc herniation which was treated with manual therapy
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
In a study that was approved nine years ago (EK-22/2009) we could show (i) that spinal manipulative therapy (SMT) is a very effective and safe treatment for acute and chronic lumbar disc herniation (LDH); (ii) that SMT is as effective and less expensive than lumbar nerve root injections and (iii) that the recurrence rate up to one year was very low in acute and in chronic LDH patients. However, the long-term outcome of this conservatively treated LDH patients is unknown. Thus, the objective of this amendment is to investigate the proportion of long-term recurrences in these patients who were treated with SMT for their LDH and to compare these results with already existing data from other treatments, e.g. surgery. This is important information to know whether this conservative method is a sustainable approach for treating LDH.

DETAILED DESCRIPTION:
All 148 patients with magnetic resonance imaging-confirmed disc herniation who were recruited for the study EK 22-2009 will be re-contacted to assess the course of their back problem during the past approx. nine years using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

-The same patients who were recruited for the study EK-22/2009

Exclusion Criteria:

* The same as for study EK-22/2009:

Patients with specific pathologies of the lumbar spine that are contraindications to chiropractic manipulative treatment, such as tumors, infections, inflammatory spondylarthropathies, acute fractures, Paget's disease and severe osteoporosis, will be excluded. Also excluded will be patients with previous spinal surgery, signs of cauda equina syndrome (CES), sequestration of disc material, body mass index >30, spondylolisthesis, neurogenic claudication and pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The same patients who were recruited for the study EK-22/2009: Patients with lumbar disc herniation that is treated with spinal manipulation
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
intensity of low back pain | 1 month
  intensity of low back pain in the last month (numeric rating scale)

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Mayr, M Chiro Med, Principal Investigator — Universitätsklinik Balgrist
Locations (1):
- Chiropraktik am Schaffhauserplatz, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No